CLINICAL TRIAL: NCT01576367
Title: An Open-label Extension Study to Assess Efficacy, Safety and Tolerability of Canakinumab and the Efficacy and Safety of Childhood Vaccinations in Patients With Cryopyrin Associated Periodic Syndromes (CAPS)
Brief Title: Efficacy, Safety and Tolerability of ACZ885 in Pediatric Patients With the Following Cryopyrin-associated Periodic Syndromes: Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome, or Neonatal Onset Multisystem Inflammatory Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: CACZ885D2307E1; 2011-005154-57 (EudraCT Number)
Record Dates: First submitted 2012-02-17; First posted 2012-04-12 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Cryopyrin-associated Periodic Syndromes; Familial Cold Autoinflammatory Syndrome; Muckle-Wells Syndrome; Neonatal Onset Multisystem Inflammatory Disease
Keywords: Cryopyrin-associated periodic syndromes (CAPS); Familial Cold Autoinflammatory Syndrome (FCAS); Muckle-Wells Syndrome (MWS); Neonatal Onset Multisystem Inflammatory Disease (NOMID); children, systemic autoinflammatory disease; CIAS-1 gene; NALP-3; NLRP3; ACZ885; canakinumab; human monoclonal anti-human interleukin-1 antibody; autosomal dominant; familial autoinflammatory syndrome; childhood immunizations vaccinations
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- canakinumab (Experimental): Patients will receive a standard dose at an equivalent of 2 mg/kg s.c. of canakinumab (ACZ885) every 8 weeks. Possible dose and/or dosing regimen adjustments that can be administered include: 4 mg/kg s.c. (every 4 to 8 weeks) 6 mg/kg s.c. (every 4 to 8 weeks) 8 mg/kg s.c. (every 4 to 8 weeks)
  Interventions: Biological: ACZ885

INTERVENTIONS:
Biological: ACZ885
  Other Names: Canakinumab

SUMMARY:
This trial will provide long-term safety, efficacy and tolerability of ACZ885 in CAPS patients that completed the CACZ885D2307 study

ELIGIBILITY:
Inclusion criteria:

1. Patients who completed the core CACZ885D2307 study (a patient is defined as having completed the core study if they completed the study up to and including the EOS visit with no major protocol deviations in the core).
2. Male and female patients that are ≥ 1 year of age at the time of the roll-over visit.
3. Parent or legal guardian written informed consent must be obtained before any assessment in the extension CACZ885D2307E1 study is performed.

Exclusion criteria:

1. Patients for who continued treatment in the CACZ885D2307E1 extension study is not considered appropriate by the treating physician.
2. Patients who discontinued from the core CACZ885D2307 study

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2015-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Laken
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Le Kremlin-Bicêtre, France
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Saint Augustin
  - Novartis Investigative Site, Tübingen
- Spain (2):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Lausanne, Switzerland
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Brogan PA, Hofer M, Kuemmerle-Deschner JB, Kone-Paut I, Roesler J, Kallinich T, Horneff G, Calvo Penades I, Sevilla-Perez B, Goffin L, Lauwerys BR, Lachmann HJ, Uziel Y, Wei X, Laxer RM. Rapid and Sustained Long-Term Efficacy and Safety of Canakinumab in Patients With Cryopyrin-Associated Periodic Syndrome Ages Five Years and Younger. Arthritis Rheumatol. 2019 Nov;71(11):1955-1963. doi: 10.1002/art.41004. Epub 2019 Sep 9. PMID 31161734

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Canakinumab
Started | 17
Completed | 14
Not Completed | 3
Not completed — Unsatisfactory therapeutic effect | 2
Not completed — Moved to commercial use after 6 months | 1

BASELINE CHARACTERISTICS:
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age at start of extension study (years) | 3.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Without Disease Relapse as Determined by the Physician's Global Assessment of Autoinflammatory Disease Activity, Assessment of Skin Disease and Serological Inflammation Markers.
Description: Disease relapse following complete response is defined as inflammation markers: C-Reactive Protein (CRP) and/or Serum Amyloid A (SAA) result > 30 mg/L AND Physician's Global Assessment of Autoinflammatory Disease Activity > minimal or Physician's Global Assessment >= minimal AND Skin Disease Assessment > minimal. Physician's Global Assessment of Autoinflammatory Disease Activity and Skin Disease Assessment (urticarial skin rash) are completed by the investigator using a 5 point rating scale: absent, minimal, mild, moderate and severe.
Time Frame: Week /80, 104, 128, and 152 (A minimum of 6 months and maximum of 24 months)
Population: Extension Full analysis set (FAS) consisted of all patients who received at least one dose of study drug in the extension study
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Percentage of participants | 94.1

2. Secondary Outcome: Immunogenicity of Canakinumab (ACZ885). Number of Participants With Anti-canakinumab Antibodies
Description: Immunogenicity assessment included determination of anti-canakinumab (ACZ885) antibodies in serum samples using BIAcore system, with detection based on surface plasmon resonance technique.
Time Frame: minimum of 6 months and maximum of 24 months
Population: Extension Safety set consisted of all patients from the core study who received at least one dose of study drug in the extension study and had at least one post-treatment safety assessment. Of note, the statement that a patient had no AE also constituted a safety assessment.
Measure: Number; unit: Participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Change From Baseline (Core Study Baseline) in C--Reactive Protein (CRP) and Serum Amyloid A (SAA) Concentrations
Description: CRP and SAA were used as serologic inflammatory markers. The target level concentrations for CRP and SAA was ≤15 mg/L and ≤10 mg/L, respectively. Negative change in concentration of inflammatory markers indicated improvement.
Time Frame: Week 0, 80, 104, 128 and 152, last assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (mg/L)
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
(mg/L)
  CRP at Core End of Study (last assessment) (n=14) | -5.4 (6.28)
  CRP at week 80 (n=16) | -14.7 (35.8)
  CRP at Week 104 (n=11) | -3.8 (14.4)
  CRP at Week 128(n=12) | -4.1 (10.3)
  CRP at Week 152 (n=12) | -4.3 (11)
  CRP at End of Study (last assessment) (n=16) | -10.4 (30.3)
  SAA at Core End of Study (last assessment) (n=16) | -54.4 (133.8)
  SAA at Week 80 (n=12) | -79.1 (224.1)
  SAA at week 104 (n=11) | 15.8 (158.1)
  SAA at week 128 (n=10) | -28.2 (47.4)
  SAA at week 152 (n=11) | -6.4 (60.0)
  SAA at End of Study (last assessment) (n=15) | -58.5 (183.6)

4. Secondary Outcome: Frequency Counts of Physician's Global Assessment of Autoinflammatory Disease and Skin Disease
Description: Participants were assessed based by physician on Physician's Global Assessment measured on a 5--point scale for auto inflammatory disease activity as: 0 = None/absent; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe
Time Frame: minimum of 6 months and maximum of 24 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Percentage of participants
  Assessment of autoinflammatory disease (Absent) | 64.7
  Assessment of autoinflammatory disease (Minimal) | 29.4
  Assessment of autoinflammatory disease (Mild) | 5.9
  Assessment of autoinflammatory disease (Moderate) | 0
  Assessment of autoinflammatory disease (Severe) | 0
  Assessment of skin disease (Absent) | 94.1
  Assessment of skin disease (Minimal) | 0
  Assessment of skin disease (Mild) | 5.9
  Assessment of skin disease (Moderate) | 0
  Assessment of skin disease (Severe) | 0

5. Secondary Outcome: Number of Vaccination Cases With Protective Antibody Levels Following Immunization With Inactivated Vaccines
Description: Participants who received any inactivated vaccines during the study were assessed for their ability to attain protective antibody levels against the vaccine (antigen) post immunization. Participants vaccinations were not assessed for a response if the antibody titre was already sufficient at pre-dose and maintained during the study.
Time Frame: pre-vaccine dose, Day 28 post-vaccine
Population: Extension Full analysis set (FAS) consisted of all patients who received at least one dose of study drug in the extension study. Out of 20 unique patient-vaccination cases, 17 cases were assessable for a vaccination response due to availability of pre dose antibody titer.
Measure: Number; unit: vaccination cases
Units Other Than Participants: patient-vaccination cases
Arm/Group | Canakinumab
Number analyzed (Participants) | 4
Number analyzed (patient-vaccination cases) | 17
vaccination cases
  Positive response for antibody levels | 16
  No pre-dose antibody levels | 3

ADVERSE EVENTS:
Arm/Group | Canakinumab
Serious Adverse Events (participants affected / at risk) | 8/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=17)
Conductive deafness (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Papillitis (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Limb injury (Injury, poisoning and procedural complications) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=17)
Eosinophilia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cryopyrin associated periodic syndrome (Congenital, familial and genetic disorders) | 1
Conductive deafness (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Eye pruritus (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 1
Papilloedema (Eye disorders) | 2
Uveitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Gingival hypertrophy (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Pyrexia (General disorders) | 6
Milk allergy (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Abscess limb (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 3
Eczema infected (Infections and infestations) | 1
Enterobiasis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Hand-foot-and-mouth disease (Infections and infestations) | 1
Impetigo (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Lice infestation (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 2
Varicella (Infections and infestations) | 3
Vulval abscess (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Body temperature increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
CSF white blood cell count increased (Investigations) | 1
Serum amyloid A protein increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Tympanometry abnormal (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Burning sensation (Nervous system disorders) | 1
Cerebral ventricle dilatation (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hemiplegia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Motor developmental delay (Nervous system disorders) | 2
Pyramidal tract syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Speech disorder developmental (Nervous system disorders) | 3
Hypertonic bladder (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.